CLINICAL TRIAL: NCT01033903
Title: Which is the Optimal Treatment for Miscarriage With a Gestational ac in the Uterus and Which Factors Can Predict if the Treatment Will be Successful?
Brief Title: Optimal Treatment of Miscarriage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2007-007661-20
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Abortion, Spontaneous
Keywords: Abortion, Spontaneous; Randomized Controlled Trial
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol 800 micrograms intravaginally (Experimental)
  Interventions: Drug: misoprostol
- expectant managment (No Intervention)

INTERVENTIONS:
Drug: misoprostol — 800 micrograms intravaginally ONCE
  Arms: Misoprostol 800 micrograms intravaginally

SUMMARY:
The main objective of the study is to determine if there is a difference in the number of women with a complete miscarriage after 10 days between expectant management versus treatment with 800 micrograms of misoprostol intravaginally in women with an an incomplete miscarriage before 14 weeks and a gestational sac retained in the uterus.

ELIGIBILITY:
Inclusion Criteria:

* nonviable intrauterine pregnancy with retained gestational sac in the uterus
* the embryo if visible 5 to 35 mm without a heart beat
* vaginal bleeding
* circulatory stable
* hemoglobin at least 80 g/L

Exclusion Criteria:

* contraindications against misoprostol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2008-10-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
complete miscarriage | 10 days

SECONDARY OUTCOMES:
complete miscarriage | 17 days, 24 days, 31 days

CONTACTS AND LOCATIONS:
Locations (1):
- Region Skane, Kvinnokliniken, University Hopsital MAS, Malmo, Sweden

REFERENCES:
- [Derived] Fernlund A, Jokubkiene L, Sladkevicius P, Valentin L. Misoprostol treatment vs expectant management in women with early non-viable pregnancy and vaginal bleeding: a pragmatic randomized controlled trial. Ultrasound Obstet Gynecol. 2018 Jan;51(1):24-32. doi: 10.1002/uog.18940. Epub 2017 Dec 5. PMID 29072372